CLINICAL TRIAL: NCT03003377
Title: Comparison of the Sevoflurane EC50 Values for Laryngeal Mask Airway Supreme Versus Laryngeal Mask Airway ProSeal Insertion During Target-controlled Infusion of Remifentanil. A Randomized Trial
Brief Title: Sevoflurane-remifentanil EC50 (The 50% Effective Concentration) Values for LMA-Supreme Versus LMA ProSeal Insertion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Matilde Zaballos, Clinical professor, Hospital General Universitario Gregorio Marañon
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CETSEVOREM
Record Dates: First submitted 2016-11-15; First posted 2016-12-28 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Sevoflurane
Keywords: Sevoflurane; Remifentanil; Laryngeal mask supreme; laryngeal mask proseal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Device: laryngeal mask supreme (Experimental): Determine the Sevoflurane concentration associate with remifentanil for the insertion of the laryngeal mask supreme
  Interventions: Device: laryngeal mask supreme
- Device: laryngeal mask proseal (Active Comparator): Determine the Sevoflurane concentration associate with remifentanil for insertion of the laryngeal mask ProSeal
  Interventions: Device: laryngeal mask proseal

INTERVENTIONS:
Device: laryngeal mask supreme — Sevoflurane was administered by facial mask with concomitant remifentanil administration (at an effect-site of 4 ng/ml). The LMAS was inserted according to the manufacturer's recommendations with the patient's head in the neutral position. After equilibrium the LMAS was inserted and secured according to the manufacturer's recommendations, without using muscle relaxants. A single measurement will be obtained from each patient. If the patient reacted with movement, a 1-2 mg/kg dose of Propofol was administered.
  Arms: Device: laryngeal mask supreme
Device: laryngeal mask proseal — Sevoflurane was administered by facial mask with concomitant remifentanil administration (at an effect-site of 4 ng/ml).The LMAP was inserted according to the manufacturer's recommendations with the patient's head in the neutral position. After equilibrium the LMAP was inserted and secured according to the manufacturer's recommendations, without using muscle relaxants. A single measurement will be obtained from each patient. If the patient reacted with movement, a 1-2 mg/kg dose of Propofol was administered.
  Arms: Device: laryngeal mask proseal

SUMMARY:
The study was designed to determine and compare the sevoflurane EC50 optimal concentration for laryngeal mask airway Supreme versus laryngeal mask airway ProSeal insertion during target-controlled infusion of remifentanil.

DETAILED DESCRIPTION:
Since the introduction of the laryngeal mask airway (LMA), a number of new supraglottic airway devices as the LMA-Supreme (LMAS) and the LMA ProSeal (LMAP) have been developed for the management of the airway during general anesthesia, and specifically in the context of day surgery. ProSeal laryngeal mask airway is a reusable device designed to separate the gastrointestinal and respiratory tracts, thereby improving the airway seal pressure and allowing for controlled ventilation more efficiently tan classic LMA. The LMAS was developed in 2007 as a single-use device provided with gastric canal, and combine the features of both intubating LMA and the LMAP. Recently, there has been a growing interest in these devices because of favourable studies obtained in several anaesthetic contexts that have proven their effectiveness and safety. Even though insertion of both devices were associated with a higher initial success rate, fewer airway manipulations and a safe and effective airway during anaesthesia, the anaesthetic techniques for its insertion were not standardised. Most available data on the requirements of anaesthetic drugs and co-induction agents used for insertion of both devices originate from research involving other assessments of the LMAs such as the seal respiratory and gastrointestinal tract. Investigators tested for differences in the predicted concentration of sevoflurane with remifentanil for the insertion of the LMAS vs. LMAP.

Methods: 45 patients American Society of Anesthesiologists (ASA) class I or II aged 20-60 years undergoing ambulatory elective surgery were randomized to either the LMAS or LMAP. The patients were premedicated with midazolam 1 mg iv before surgery. All patients were preoxygenated using 100% oxygen with a normal tidal volumen for 3 min. The circuit was primed with sevoflurane 5% at a fresh gas flow of 6 L/min for 1 min. Anaesthesia was induced with inhaled sevoflurane up to 5% in oxygen via facemask with fresh gas flow at 6 L/min. Simultaneously remifentanil at an effect-site of 4 ng/ml was started. Target-controlled infusions was used (Alaris PK) for remifentanil administration. After loss of consciousness, the inspired concentration of sevoflurane was changed to obtain a predetermined end-tidal concentration. A single experienced anaesthetist in the use of supraglottic devices inserted the devices according to the manufacturer's recommendations. The LMAs size was chosen according to the sex of the patients, size 4 for women and size 5 for men; however for patients weighing ≤50 kg a size 3 was inserted. Neuromuscular blocking agents were not given. Two nurses, who were blinded to the anaesthetic concentration, classified responses by the patient to LMA insertion as either "movement" or "not movement". Assesment was made for jaw relaxation and graded with Muzi score. A Muzi score >2 was defined as a failure of insertion. The end-tidal (ET) sevoflurane concentration used for each patient was determined using the Dixon's up-and-down method. The ratio of the end-tidal to predetermined end-tidal concentrations was maintained at 0.9-1.0 for at least 10 minutes to establish equilibration before device insertion was attempted. The first patient received a 2.5% sevoflurane concentration and the step size of increase/decrease was 0.5%. If the supraglottic device (LMAS or LMAP) insertion was successful, sevoflurane concentration for the next patient was decrease by 0.5%. If not, sevoflurane concentration was increased by the same amount for the next patient. For their comfort, patients experiencing movement received a 1-2 mg/kg bolus dose of propofol.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients
* Scheduled to ambulatory surgery
* Need for general anaesthesia
* General anaesthesia usually performed with laryngeal mask
* Negative pregnancy test in women
* Signed inform consent

Exclusion Criteria:

* Patients with a potentially difficult airway (Mallampati III or IV, a limited mouth opening and/or cervical spine disease)
* Patients with reactive airway disease
* Signs of upper respiratory infection
* Patients who had a risk of gastric aspiration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
To compare the the minimum alveolar anesthetic concentration (determined at 1 atmosphere, that prevents movement in 50% of patients to LMAS vs. LMAP insertion) of sevoflurane with simultaneous remifentanil infusion in adult patients. | The sevoflurane concentration is obtained during the insertion of the LMAS or LMAP in patients, after anesthesia induction
  To compare the concentration of sevoflurane with concomitant remifentanil infusion required for LMAS insertion vs. the concentration of sevoflurane with concomitant remifentanil infusion required for LMAP insertion.

SECONDARY OUTCOMES:
Blood pressure in mmHg | Baseline and every 3 minutes until 6 minutes after insertion of the LMAs
  To compare the evolution of blood pressure during insertion of LMAS group versus LMAP group
Heart rate in bpm, | Before and after LMAs insertion (every minute until 6 minutes)
  To compare the evolution of heart rate during insertion of LMAS group versus LMAP group
BIS data, number from 100 (awake) to 40-45 (anesthetic status) | Before and after LMAs insertion (every minute until 6 minutes)
  To compare the evolution of BIS values during insertion of LMAS group versus LMAP group

CONTACTS AND LOCATIONS:
Overall Officials: Maite López-Gil, MD, PhD, Study Chair — Servicio de Anestesiología, Hospital General Universitario Gregorio Marañón
Locations (1):
- Servicio de Anestesia, Hospital General Universitario Gregorio Marañón, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Monteserin-Matesanz C, Gonzalez T, Anadon-Baselga MJ, Zaballos M. Supreme laryngeal mask airway insertion requires a lower concentration of sevoflurane than ProSeal laryngeal mask airway insertion during target-controlled remifentanil infusion: a prospective randomised controlled study. BMC Anesthesiol. 2020 Jan 7;20(1):5. doi: 10.1186/s12871-019-0921-5. PMID 31910822